CLINICAL TRIAL: NCT04646252
Title: Impaired Endothelial Glycocalyx Predicts Adverse Outcome in Subjects Without Overt Cardiovascular Disease: a 6 Year Follow up Study
Brief Title: The Role of Glycocalyx Integrity in the Primary Prevention of Major Cardiovascular Events
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor, University of Athens
Other Study IDs: Glycocalyx primary prevention
Record Dates: First submitted 2020-11-22; First posted 2020-11-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Endothelial Dysfunction; Arterial Stiffness
Keywords: perfused boundary region; primary prevention of major cardiovascular events; integrity of endothelial glycocalyx

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aliquots of serum and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Perfused Boundary Region of sublingual microvessels — Measurement of Perfused Boundary Region of sublingual microvessels to assess thickness of endothelial glycocalyx Measurement of Pulse Wave Velocity to quantify arterial stiffness
  Other Names: pulse wave velocity; pulse wave analysis

SUMMARY:
The researchers intend to recruit individuals who are referred for a routine screening in the primary prevention outpatient clinic of Attikon University hospital, Athens According to institutional protocols, a detailed medical history for atherosclerotic risk factors and current medication is recorded and a baseline clinical examination is performed. Moreover fasting blood samples are drawn to diagnose the presence of diabetes mellitus and hyperlipidemia. Glycocalyx examination is performed at the same visit. The subjects are revaluated at one month and then followed up according to the attending physician's instructions. Pulse wave velocity and the rest pulse wave analysis parameters were also calculated to determine the additive predictive value for cardiovascular events beyond SCORE2. All subjects are followed up for adverse events (death, stroke, myocardial infarction, hospitalization for heart failure) for 6 years after enrollment via telephonic contact and planned appointment at the outpatient clinic.

DETAILED DESCRIPTION:
Blood pressure is measured in each subject with the aid of a digital oscillometric sphygmomanometer (TensioMed, Budapest Hungary, Ltd). Each subject rests in a quiet room at 25°C for 30 minutes before the examination. The cuff is placed in the right arm, while the subject is seated. The diagnosis of hypertension is made on the basis of:1) systolic blood pressure ≥140 mmHg/diastolic blood pressure ≥90 mmHg after 3 consecutive measurements or 2) the participant is receiving antihypertensive treatment. Moreover fasting blood samples are drawn to identify the presence of diabetes mellitus and hyperlipidemia in our sample. Specifically, DM is determined by either plasma glucose ≥ 126 mg/dl measured by the enzymatic in vitro test (Roche, automatic chemistry clinical analyzer) or treatment with antidiabetic agents . Similarly, hyperlipidemia was defined by either Total Cholesterol ≥230 mg/dl, and/or LDL ≥160 mg/dl, and /or TGs ≥200 mg /dl measured by the colorimetric spectrophotometry (Roche Diagnostics) or the use of lipid lowering agents according to the running guidelines held during the initial examination. Additionally, smokers are considered only those participants who are actively smoking at the time of enrollment . Also, the presence of positive family history of coronary artery disease is defined as coronary disease in a first degree female relative before 65 years or a male relative before 55 years of age. BMI is calculated as the ratio of weight (kg) to the square of height (m2). Furthermore, SCORE estimation system is used to calculate the 10-year cardiovascular risk for each participant.

As far as ethnicity is concerned, an individual is not considered Greek in case he/she was born abroad and also has at least a foreigner parent or he/she is born in Greece but both parents were foreigners. Inversely, a subject was considered Greek if they and simultaneously both parents were born in Greece.

Exclusion criteria are the history of Coronary artery disease (CAD), Peripheral Arterial Disease (PAD), Heart failure (HF), Stroke, hepatic or renal failure, active neoplasia and poorly controlled DM, defined as Hba1C>7%.

ENDOTHELIAL GLYCOCALYX EVALUATION The researchers quantified the perfused boundary region (PBR, measured in μm) of the sublingual microvasculature by using Sideview Darkfield Imaging (Microscan, Glycocheck, Microvascular Health Solutions Inc., Salt Lake City, UT, USA) . Briefly, SDF camera utilizes green reflected light emitting diode (LED) light (540 nm) from hemoglobin molecules to depict the radial displacements of RBCs within the microvessels . The camera is inserted under the tongue and captures more than 3000 vascular segments of vessels with diameter ranging from 5 μm to 25 μm. The images are obtained automatically by the Glycocheck software . Afterwards the system checks the quality of the recordings and selects the valid frames (contrast enhancement greater than 60%), which are going to be further analyzed . The RBC column width, as well as the total perfused diameter of microvessels is estimated by the software with high accuracy. Then PBR is calculated by the formula [Perfused Diameter- RBC column width]/2.The software also provides the PBR of vessels with diameter 5-9μm, 10-19μm, 20-25μm and the mean 5-25μm As a result, PBR expresses the outer area of the vessels' lumen that is vulnerable to RBC penetration and is consistent with the integrity of glycocalyx layer. Thus, high PBR values are considered as indicator of damaged endothelial glycocalyx with affected barrier properties, which allows high spatio-temporal distribution of RBCs. On the other hand Conversely, low PBR values are associated with robust thick glycocalyx layer. The whole procedure lasts for approximately 3 minutes, does not require high expertise, is operator independent, has satisfactory reproducibility and thus is highly recommended as a validated technique for the assessment of endothelial glycocalyx function . The PBR measurements are independent of red blood cell filling of the vessels segments (hematocrit), because the software only includes vessel segments that have a filling percentage of more than 50%. Hence, vessel segments are only selected when at least 11 of the 21-line markers have a positive signal for the presence of an erythrocyte. Thus, PBR values are independent of hematocrit, reflecting a damaged glycocalyx that is more accessible for circulating erythrocytes .

In the current study the evaluation of PBR takes place between 9:00 and 11:00, after 8 hours fasting and abstinence from alcohol and smoking and temporary discontinuation of medications for 48 h before the examination as well.

PULSE WAVE VELOCITY Pulse wave velocity carotid to femoral and Augmentation Index were estimated non-invasively using a dedicated technique (Complior, Alam Medical, Vincennes, France).

FOLLOW UP A follow up assessment is performed 6 years after the recruitment via telephonic contact and planned appointment at the outpatient clinic. Briefly, at the reevaluation the participants or their legal representatives - in case of inability or death- are asked for the incidence of major cardiovascular events or death attributed to any cause. The primary composite outcome of major adverse events consists of death, myocardial infarction (ICD-10: DI20-22), stroke (ICD-10: DI60-68; DG45) and hospitalization for heart failure (ICD-10: DI50-51; DI42; DI11). Each of the forenamed events is documented by hospital medical records or attending phycians' letters and confirmed by the national security electronic records using the appropriate ICD10.

STATISTICAL ANALYSIS

Statistical analysis is performed by SPSS version 25 (IBM SPSS Statistics, Inc., Chicago, IL) and Stata version 16 (StataCorp LP, College Station, TX). Scale variables are presented as mean ±SD in case of normal distribution, as determined by the normality tests Kolmogorov-Smirnov test and Shapiro-Wilk, or as medians and interquartile ranges in case of non-normal distribution. Nominal variables are expressed as frequencies and percentages. Scale variables are compared using independent samples Student's t tests or Mann-Whitney tests as indicated, whereas categorical variables are compared using Chi-square tests or Fisher's exact tests, as appropriate. In addition, patients are dichotomized based on the mean values of PBR for the sublingual microvessel diameter 5-25μm, 5-9 μm, 10-19 μm, and 20-25 μm . Cox proportional hazard models are built for each variable to decide whether any of mean values of the above PBR categories can serve as an independent predictor of major cardiovascular events or death at a significance level of p value<0.05. Cumulative event rates are calculated using the Kaplan-Meier survival analysis for subjects with lower vs higher mean PBR value. The log-rank test for time-to-event data with respect to the total events is used for comparison of these two groups. Cox proportional hazard models are built for each possible risk factor in relation to the study endpoints. Estimated hazard ratios and their respective 95% confidence intervals are obtained. P value<0.05 are considered significant. Multivariate analysis include factors with proven clinical value or p value ≤0.1 at univariate analysis. Moreover, chi-square values of multivariate models were comparedbefore and after adjusting for PBR. Chi square change with p value<0.05 is considered significant. Furthermore, the net reclassification index (NRI) and Harrell's C were calculated to evaluate improvement in risk prediction by PBR and p value<0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

We recruit individuals who were referred for a routine screening in the primary prevention outpatient clinic of Attikon University hospital.

Exclusion Criteria:

* History of Coronary artery disease,
* History of Peripheral Arterial Disease,
* History of Heart failure
* History of Stroke
* hepatic failure
* renal failure,
* active neoplasia
* poorly controlled DM, defined as Hba1C>7%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As far as ethnicity is concerned, an individual is not considered Greek in case he/she was born abroad and also has at least a foreigner parent or he/she is born in Greece but both parents were foreigners. Inversely, a subject was considered Greek if they and simultaneously both parents were born in Greece..
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-01-10 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular events | 6 years
  death of any cause, myocardial infarction (ICD-10: DI20-22), stroke (ICD-10: DI60-68; DG45) and hospitalization for heart failure (ICD-10: DI50-51; DI42; DI11).

CONTACTS AND LOCATIONS:
Overall Officials: IGNATIOS IKONOMIDIS, PROFESSOR, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

REFERENCES:
- [Derived] Ikonomidis I, Thymis J, Simitsis P, Koliou GA, Katsanos S, Triantafyllou C, Kousathana F, Pavlidis G, Kountouri A, Polyzogopoulou E, Katogiannis K, Vlastos D, Kostelli G, Triantafyllidi H, Parissis J, Papadavid E, Lekakis J, Filippatos G, Lambadiari V. Impaired Endothelial Glycocalyx Predicts Adverse Outcome in Subjects Without Overt Cardiovascular Disease: a 6-Year Follow-up Study. J Cardiovasc Transl Res. 2022 Aug;15(4):890-902. doi: 10.1007/s12265-021-10180-2. Epub 2021 Oct 28. PMID 34713396